CLINICAL TRIAL: NCT03309813
Title: A Feasibility Study of Focused Ultrasound to Perform Bilateral Medial Thalamotomy for the Treatment of Chronic Trigeminal Neuropathic Pain
Brief Title: Feasibility Study of ExAblate Thalamotomy for Treatment of Chronic Trigeminal Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP002
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-12

CONDITIONS: Trigeminal Neuropathic Pain
Keywords: ExAblate; TcMRgFUS; Thalamotomy

STUDY DESIGN:
Intervention Model Description: Subjects were randomized to an Exablate Test Arm or a Sham Control Arm. After completing the Month 3 Sham study visit, Sham Controls could elect to receive the actual Exablate ablation (same as test arm) and continue follow-up in a "Crossover Arm."
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial ExAblate (Experimental): ExAblate Transcranial MR Guided Focused Ultrasound (MRgFUS)
  Interventions: Device: Transcranial ExAblate
- Sham Transcranial ExAblate (Sham Comparator): ExAblate MRgFUS Sham Procedure
  Interventions: Device: Sham Transcranial ExAblate; Device: Crossover Transcranial Exablate

INTERVENTIONS:
Device: Transcranial ExAblate — ExAblate Thalamotomy for Chronic Trigeminal Neuropathic Pain
  Other Names: MRgFUS; Thalamotomy
  Arms: Transcranial ExAblate
Device: Sham Transcranial ExAblate — Sham ExAblate Thalamotomy procedure
  Arms: Sham Transcranial ExAblate
Device: Crossover Transcranial Exablate — Subjects randomized to the Sham Exablate could opt for the Crossovover Transcranial Exablate Arm (Exablate Thalamotomy) after completing the Month 3 visit in the Sham Arm.
  Other Names: MRgFUS; Thalamotomy
  Arms: Sham Transcranial ExAblate

SUMMARY:
The goal of this prospective, randomized, sham-controlled, crossover study is to evaluate the safety and feasibility of ExAblate Neuro treatment of chronic trigeminal neuropathic pain.

DETAILED DESCRIPTION:
This study is to show that for patients with treatment-refractory chronic trigeminal neuropathic pain, ExAblate Neuro focused ultrasound (FUS) can safely create lesions bilaterally in the thalamic nuclei to reduce pain and provide functional benefits in daily activities. After informed consent and screening, eligible subjects will be randomized to either an ExAblate treatment or a Sham Control procedure. Subjects who are randomized to Sham Control will undergo the same procedure and follow-up visits through their Month 3 visit. After the Month 3 assessments are complete, all subjects will be un-blinded and those in the Sham treated group will have the option for an actual ExAblate treatment in an un-blinded fashion, as long as they still qualify for ExAblate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 18 and 75 years, inclusive
* Subjects who are able and willing to give consent and able to attend all study visits
* Severe chronic, trigeminal neuropathic pain of ≥6 months duration.
* Pain is medication-refractory to adequate trials of at least 3 prescription medications commonly used for symptomatic relief of neuropathic pain with current adjunctive use of at least one medication. An adequate medication trial is defined as a therapeutic dose of each medication without sufficient effect.
* Pain is treatment-resistant to at least one interventional therapies including injections, procedures, neuromodulation, and surgery.
* Able to communicate sensations during the focused ultrasound treatment
* Stable prescribed doses of all symptomatic pain medications for 30 days prior to study entry and for the duration of the 3-month blinded phase of the study.

Exclusion Criteria:

* Craniofacial pain syndromes related to malignancy of the head and neck
* Idiopathic trigeminal neuralgia
* Headache syndromes like migraine, cluster headache
* Temporomandibular joint syndrome
* Atypical facial pain or pain related to a somatoform disorder
* Subjects with active psychiatric illness will be excluded. For the purpose of this study, active psychiatric illness includes:

  * Exhibiting current suicide ideation and/or a history of suicide attempt within past 2 years
  * been hospitalized for the treatment of a psychiatric illness within the past 2 years
  * received transcranial magnetic stimulation for depression treatment
  * received electroconvulsive therapy for depression
* Any presence or history of psychosis will be excluded.
* Subjects with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Subjects with documented myocardial infarction within six months of protocol entry
  * Significant congestive heart failure defined with ejection fraction < 40
  * Subjects with unstable ventricular arrhythmias
  * Subjects with atrial arrhythmias that are not rate-controlled
* Severe hypertension (diastolic BP > 100 on medication)
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hours of total table time.)
* Subjects participating or have participated in another clinical trial in the last 30 days
* Presence of systemic neurological disease or dysfunction
* Known life-threatening systemic disease
* Subjects with brain tumors or any significant intracranial mass. Trigeminal or cavernous sinus tumors causing neuropathic pain are not excluded.
* Pregnancy or lactation
* Legal incapacity or limited legal capacity
* Subjects with a deep brain stimulation implant or with a prior stereotactic thalamic ablation
* History of hemorrhagic stroke or cerebrovascular event within the past year of treatment exhibiting incomplete resolution
* History of seizures within past year of treatment
* Severe kidney disease or on dialysis
* Subjects who are unable to tolerate medications due to intolerable side effects.
* Subjects with pain other than craniofacial neuropathic pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William J Elias, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Ishaque M, Moosa S, Urban L, Kundu B, Qureshi Z, Spears T, Fletcher PT, Donahue J, Patel SH, Goldstein RB, Finan PH, Liu CC, Elias WJ. Bilateral focused ultrasound medial thalamotomies for trigeminal neuropathic pain: a randomized controlled study. J Neurosurg. 2023 Dec 29;140(6):1799-1809. doi: 10.3171/2023.10.JNS23661. Print 2024 Jun 1. PMID 38157521

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial ExAblate (MRgFUS) Only: ExAblate Transcranial MR Guided Focused Ultrasound (MRgFUS)
  Transcranial ExAblate: ExAblate Thalamotomy for Chronic Trigeminal Neuropathic Pain
- Sham Transcranial ExAblate First, Then Optional Transcranial Exablate (MRgFUS): ExAblate MRgFUS Sham Procedure
  Sham Transcranial ExAblate: Sham ExAblate Thalamotomy procedure
Period: Main Randomized Study
Arm/Group | Transcranial ExAblate (MRgFUS) Only | Sham Transcranial ExAblate First, Then Optional Transcranial Exablate (MRgFUS)
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Crossover Transcranial Exablate
Arm/Group | Transcranial ExAblate (MRgFUS) Only | Sham Transcranial ExAblate First, Then Optional Transcranial Exablate (MRgFUS)
Started (Subjects randomized to Sham Transcranial Exablate (n=5) were given the option to receive the Exablate treatment and follow up in the Crossover Exablate group. Thus, the number of subjects participating in the Crossover Exablate group may not equal the number of subjects completing the Sham group 3 Month visit.) | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Transcranial ExAblate First, Then Optional Transcranial ExAblate (MRgFUS): ExAblate MRgFUS Sham Procedure
  Sham Transcranial ExAblate: Sham ExAblate Thalamotomy procedure
  Crossover Transcranial Exablate: Subjects randomized to the Sham Exablate could opt for the Crossovover Transcranial Exablate Arm (Exablate Thalamotomy) after completing the Month 3 visit in the Sham Arm.
- Total: Total of all reporting groups
Arm/Group | Transcranial ExAblate (MRgFUS) Only | Sham Transcranial ExAblate First, Then Optional Transcranial ExAblate (MRgFUS) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 64.3 (8.9) | 59.6 (7.9) | 62.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Severity of Device and Procedure Related Complications
Description: To evaluate the incidence and severity of adverse events associated with ExAblate lesioning of the bilateral medial thalamus for painful neuropathies of the face and head that are severe and treatment-refractory.
Time Frame: At the time of ExAblate Transcranial thalamotomy procedure through 3-months post-thalamotomy
Reporting Status: Not Posted, anticipated posting 2023-10

2. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Numeric Pain Rating Scale (NPRS) change in worst pain experienced over 24 hours before and at 3 months following bilateral FUS medial thalamotomy versus sham procedures was determined from the 11-point numeric pain rating scale with 0 as no pain and 10 the worst pain imaginable. High NPRS scores are worse pain (0 is no pain, 10 is maximum). Percent change from Baseline at Month 3 was calculated as follows: 100*(NPRS Score at Baseline - NPRS Score at Month 3)/NPRS Score at Baseline. High percent change in NPRS Score from Baseline is better (improved pain).
Time Frame: Percent Change in NPRS from before treatment to 3 Months following treatment.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Sham Transcranial ExAblate First: ExAblate MRgFUS Sham Procedure
  Sham Transcranial ExAblate: Sham ExAblate Thalamotomy procedure
- Optional Crossover Transcranial Exablate (MRgFUS): After completing the 3 Month Visit sham subjects were given the opportunity to receive the Exablate treatment and continue follow-up in the Crossover Group.
Arm/Group | Transcranial ExAblate (MRgFUS) Only | Sham Transcranial ExAblate First | Optional Crossover Transcranial Exablate (MRgFUS)
Number analyzed (Participants) | 5 | 5 | 3
Percent change | -9.7 (27.4) | 12.9 (21.7) | 4.8 (8.3)

3. Secondary Outcome: Pain Interference Scale 8a v1.0 From the Patient-Reported Outcomes Measurement Information Systems (PROMIS) Pain Inventory
Description: The Pain Interference 8a v1.0 Scale (Short Form) from the Patient-Reported Outcomes Measurement Information Systems (PROMIS) Pain Inventory is an 8-item patient completed short form with each item on a 5-point scale (0-4). The total score possible ranges from 0-32. The PROMIS pain interference scale measures the degree to which pain interferes with activities of daily living. A high percent change from Baseline at 3 Months post-treatment is better, shows improvement.
Time Frame: From pre-treatment through 3 months following treatment.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- CrossoverTranscranial Exablate: After completing the 3 Month Visit sham subjects were given the opportunity to receive the Exablate treatment and continue follow-up in the Crossover Group.
Arm/Group | Transcranial ExAblate | Sham Transcranial ExAblate | CrossoverTranscranial Exablate
Number analyzed (Participants) | 5 | 5 | 3
Percent Change | 12.9 (28.3) | 16.6 (30.5) | 54.7 (40.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected though 3 months post-thalamotomy.
Groups:
- Transcranial ExAblate (MRgFUS): ExAblate Transcranial MR Guided Focused Ultrasound (MRgFUS)
  Transcranial ExAblate: ExAblate Thalamotomy for Chronic Trigeminal Neuropathic Pain
Arm/Group | Transcranial ExAblate (MRgFUS) | Sham Transcranial ExAblate First | Optional Crossover Transcranial Exablate (MRgFUS)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial ExAblate (MRgFUS) (N=5) | Sham Transcranial ExAblate First (N=5) | Optional Crossover Transcranial Exablate (MRgFUS) (N=3)
Worsening pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Worsening pain. The subject in the sham group experienced worsening facial pain due to progression of neuropathic pain.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial ExAblate (MRgFUS) (N=5) | Sham Transcranial ExAblate First (N=5) | Optional Crossover Transcranial Exablate (MRgFUS) (N=3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) — Procedure related
Sleepiness (General disorders) | 1 (1) | 0 (0) | 0 (0) — Procedure related
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) — Procedure related
Cold sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) — Transient pain/discomfort, resolved within 72 hours.
Sonication pain (General disorders) | 1 (1) | 0 (0) | 1 (1) — Transient pain/discomfort, resolved within 72 hours.
Unsteadiness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Procedure related
Tight sensation (General disorders) | 1 (1) | 0 (0) | 0 (0) — Transient pain/discomfort, resolved within 72 hours
Facial edema (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Stereotactic frame related
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Numbness/tingling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Transient headache (General disorders) | 0 (0) | 2 (2) | 0 (0) — Transient, resolved within 72 hours
Head pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Stereotactic frame related
Pin site pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Stereotactic frame related

LIMITATIONS AND CAVEATS:
This is a pilot study with limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03309813/Prot_001.pdf